

# VALUES AND VIRTUES OF GRANDPARENTS CARING FOR THEIR GRANDCHILDREN AS PROTECTIVE FACTORS OF THEIR HEALTH AND PSYCHOLOGICAL WELLBEING



# PATIENT INFORMATION DOCUMENT AND INFORMED CONSENT

Clinical study "PSYCHO-EDUCATIONAL INTERVENTION ON STRENGTHS AND EMOTIONAL COMPETENCES TO IMPROVE PSYCHOLOGICAL WELL-BEING AND QUALITY OF LIFE IN GRANDPARENT CAREGIVERS" associated with the research project "VALUES AND VIRTUES OF GRANDPARENTS AS PROTECTIVE FACTORS OF HEALTH AND PSYCHOLOGICAL WELL-BEING".

# 1) Information to the patient about the object of the study:

Recent sociodemographic changes have resulted in greater involvement of grandparents in the upbringing and education of their grandchildren, becoming key figures of instrumental, emotional and economic support. An increasing number of grandparents are caring for their grandchildren on a regular basis, with the percentage of Spanish grandparents being the second highest in Europe.

Despite these data, studies in this area are still scarce and, moreover, have focused mainly on the negative aspects of caregiving. However, recent studies have found positive consequences of caring for grandchildren for grandparents' health and life satisfaction, finding differences not so much in terms of the number of hours the grandparents care for their grandchildren, but rather in terms of the resources and emotional competences they have.

Likewise, intervention programs with grandparent caregivers have focused on softening the negative impact of caregiving, with a tendency to focus on the grandparents' protective factors and strengths. In this line, this project will develop an intervention program based on protective factors (strengths and emotional competences), with which to enhance the psychological well-being and quality of life of grandparent caregivers.



### What does your participation consist of?

To participate in this study you must have at least 1 grandchild under 18 years of age.

We request your informed consent to authorize us to:

- Collect clinical data in coded form, in a database located at the CEU-San Pablo University in which your name will not appear and will be used exclusively for research purposes.
- Carry out a psycho-educational therapy intervention in which tools will be provided to develop
  their strengths and emotional competences. The intervention will include 5 sessions of 90
  minutes, with one week between sessions. It is a group intervention in which between 4 and 6
  grandparents will participate, in order to generate a space for exchange and share practical
  strategies. The following topics will be addressed: the role of grandparents, limits in the
  caregiving function, personal safety as a caregiver, emotional self-regulation and family
  communication.
- People who are on the waiting list can also choose to answer the questionnaires to be part of
  the control group (group that does not receive intervention), to find out if there is a difference
  between participating or not participating in the intervention. The latter will not preclude them
  from participating in an intervention at a later date.
- Administer a series of questionnaires before and after the intervention with the objective of finding out the variables associated with the grandparents' psychological well-being and quality of life. Three months after the intervention, the questionnaires would be administered again to find out if the results obtained are maintained over time. These questionnaires will ask about aspects related to the following variables: character strengths, overload, role satisfaction, emotional competences, quality of life and psychological well-being, as well as sociodemographic variables and relationship with the grandchild. The questionnaire will be completed online through the Microsoft Forms platform. It will take approximately 30 minutes to complete the form.
- In case you decide to participate, you should know that you can withdraw from the research at any time without having to give explanations. In the event that you wish to exercise your rights of access, rectification, opposition and cancellation, your data will be deleted from the file. In addition, the processing of your data will be discontinued.



### What are the benefits of participating in the study?

Participation in this study will allow you, first of all, to learn about your psychological strengths and emotional competences in relation to caring for your grandchildren. It is also expected that participating in the psychoeducational intervention will provide you with tools that will promote a more satisfying relationship with your grandchildren, as well as enhance your psychological well-being and quality of life.

### What are the risks of participating in the study?

Participation in this study is risk-free for participants and participation is completely voluntary. If at any time during the data collection or the intervention you feel uncomfortable, you can stop answering and your data will not be collected.

If you have any questions, please contact Dra. Cristina Noriega García (cristina.noriegagarcia@ceu.es) at her e-mail address where you can make any inquiry.

## 2) Informed consent:

- 1. I have read and understood the information sheet of the study.
- 2. I have had the opportunity to ask questions.
- 3. My questions have been answered to my satisfaction.
- 4. I have received sufficient information about the study and the tests to be performed.
- 5. I understand that participation is voluntary and I may discontinue my participation during the completion of the required questionnaires at any time.
- 6. In accordance with the provisions of Regulation (EU) 2016/679 of the European Parliament and of the Council of 27 April 2016 on the protection of natural persons with regard to the processing of personal data and on the free movement of such data and repealing Directive 95/46/EC, as well as other current and applicable regulations on the protection of personal data, I have been informed that my personal data, obtained through the completion of this



form as well as those resulting from my participation in the project will be processed under the responsibility of the SAN PABLO CEU UNIVERSITY FOUNDATION (hereinafter, FUSP-CEU), in order to manage my participation in this research project. In addition, I have been informed of the following aspects:

- a. That profiling is planned for the purpose of analyzing or predicting aspects of my health.
- b. That the indicated treatments are legitimized by the consent given by me.
- c. That my personal data, obtained through the completion of this form, as well as those resulting from my participation in the project will be kept for the time necessary for the development of this research, which is estimated to be 3 years, being subsequently destroyed, without being able to be kept without having been previously pseudo-anonymized. In any case, they cannot be transferred without my express consent and I do not give it in this act.
- d. That I can contact the Data Protection Delegate of FUSP-CEU, by sending my request in writing to the postal address C/ Tutor nº 35 28008 Madrid or to the e-mail address dpd@ceu.es.
- e. That in accordance with the rights conferred on me by current data protection regulations, I may contact the competent Control Authority to file the claim I deem appropriate, as well as exercise my rights of access, rectification, limitation of processing, deletion, portability and opposition to the processing of my personal data and withdraw the consent given for the processing of the same, by addressing my request to the researcher responsible at the contact address given in this document.
- 7. I agree that my written consent and other data will be made available to the clinical research project in which I am participating, and to the researchers responsible for it, Cristina Noriega García, Javier López Martínez and Leyre Galarraga Cristóbal, but always respecting confidentiality and the guarantee that my data will not be publicly available so that I can be identified.
- 8. The data collected for this study will be included, with those of other persons participating in this study, in a personal database of the CEU University, to which only the researchers



approved for this project will have access, all of them being subject to the secrecy inherent to their profession or derived from a confidentiality agreement.

9. I sign this information and consent document voluntarily to express my desire to participate in this research study until I decide otherwise. By signing this consent I do not waive any of my rights. I will receive a copy of this document for my records for future reference.

| Patient's name and surname: | |
|---|---|
| ID card/Passport: | |
| <u>Signature</u> : | <u>Date</u> : |
| Name and surname of the legal re | presentative, if applicable: |
| ID card/Passport: | |
| <u>Signature</u> : | <u>Date</u> : |
| Name and surname of the researc | <u>:her</u> : Leyre Galarraga Cristóbal |
| <u>ID card</u> : 47469527B | |
| Researcher's contact address: A | v. Montepríncipe s/n. Urbanización Montepríncipe. Faculty o |
| Medicine, Department of Psychological | ogy. Pabellón MED. Office 00.22. CEU San Pablo University. 28925 |
| Alcorcón | |
| E-mail: leyre.galarragacristobal@c | ceu.es |
| <u>Phone number</u> : 680816921 | |
| Signature: | Date: 13.01.2022 |



| Vº Bº of the Study | Director | or Drincinal | Invoctigator | of the | ctudy/) |
|---|---|---|---|---|---|
| ve Be of the Study | / Director | (or Principal | investigator | or the s | stuay): |

<u>Date</u>: